CLINICAL TRIAL: NCT07393971
Title: Controller Development to Enable Individualized Assistance in Robotic Ankle Exoskeletons
Brief Title: Development of a Real-time Controller to Estimate Walking Performance Using a Bilateral Ankle Exoskeleton
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Madonna Rehabilitation Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 0587-25-FB; 55136 (Other Grant/Funding Number: Nebraska Research Initiative)
Record Dates: First submitted 2025-12-05; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-12

CONDITIONS: Healthy Young Adults
Keywords: robotic ankle exoskeleton; human-in-the-loop optimization; wearable robotics; musculoskeletal modeling; muscle activation analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single-Arm Study of a Personalized Robotic Ankle Exoskeleton Controller (Experimental): This arm employs a within-subject design with two methods of estimating metabolic cost versus the gold standard measure of metabolic cost, wherein a single participant is subjected to two distinct measurements. This design allows for a direct comparison of the effects of each method (i.e., estimation versus gold standard) within the same individual, minimizing intersubject variability and enhancing the statistical power of the analysis.
  Interventions: Device: Adaptive Torque Control System for Ankle Exoskeleton

INTERVENTIONS:
Device: Adaptive Torque Control System for Ankle Exoskeleton — This intervention uses a robotic ankle exoskeleton equipped with a real-time adaptive controller that adjusts plantarflexion torque based on each participant's walking mechanics. Unlike standard exoskeleton controllers that use fixed or pre-programmed assistance levels, this system employs human-in-the-loop optimization to continuously update torque magnitude and timing during treadmill walking. The controller integrates metabolic estimations, kinematic data, and musculoskeletal modeling to identify individualized assistance patterns that reduce walking effort and improve muscle activation efficiency. Participants complete multiple walking trials while the controller automatically modifies assistance to determine the optimal personalized settings.

SUMMARY:
This study is developing and testing a new controller for a robotic ankle exoskeleton (Biomotum) that can adjust itself in real time to better support people while they walk. The system learns how each person moves and automatically changes the amount and timing of assistance to make walking feel easier and more efficient. By using information from the person wearing the device, the exoskeleton can quickly find the level of support that works best for them. The long-term goal is to create personalized walking assistance that can help people with mobility limitations move more comfortably and with less effort.

DETAILED DESCRIPTION:
This project aims to develop and test a real-time adaptive controller for a robotic ankle exoskeleton (Biomotum) that personalizes assistance to each user by minimizing metabolic cost and optimizing muscle activation patterns during walking. Using human-in-the-loop optimization and advanced musculoskeletal modeling, the controller will dynamically adjust torque magnitude and timing to achieve optimal performance more quickly than current methods.

ELIGIBILITY:
Inclusion Criteria:

* able to walk independently on a treadmill for 10 minutes,
* free of neurological, cardiovascular, pulmonary, or musculoskeletal conditions that limit walking and exercising,
* no current lower extremity pain or injury,
* able to wear an exoskeleton and safety harness, can provide informed consent

Exclusion Criteria:

* history of neurological disease that affected gait or balance,
* current or recent lower extremity musculoskeletal injury or surgery,
* chronic lower extremity pain during walking,
* inability to participate in moderate-intensity exercise,
* require an assistive device for walking,
* any metabolic or systemic diseases that may be exacerbated by exercise

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Successful Real-Time Operation of the Robotic Ankle Exoskeleton Controller | through study completion, an average of 1 year
  Device feasibility will be evaluated by the successful real-time operation of the robotic ankle exoskeleton and adaptive controller during treadmill walking. Feasibility is defined as the controller's ability to continuously generate, update, and apply assistive torque in real time based on incoming biomechanical and physiological data without system failure, interruption, or safety-related termination. Successful operation will be confirmed by continuous controller function and synchronized data acquisition across walking trials.

SECONDARY OUTCOMES:
Net Metabolic Rate During Exoskeleton-Assisted Walking Measured by Indirect Calorimetry | through study completion, an average of 1 year
  Net oxygen consumption (VO₂) and carbon dioxide production (VCO₂) will be measured during treadmill walking using indirect calorimetry (Cosmed K5, Cosmed USA Inc., Chicago, IL). Metabolic rate will be calculated using standard equations during steady-state walking conditions. Measurements will be collected at regular intervals to characterize metabolic demand under different exoskeleton assistance configurations.
Estimated Metabolic Rate Derived From Joint-Space Musculoskeletal Modeling | through study completion, an average of 1 year
  Estimated metabolic rate will be derived from joint-space musculoskeletal models using kinematic and kinetic data collected during treadmill walking. Model-based estimates will be computed on a stride-by-stride basis to provide an indirect estimate of metabolic demand that can be compared with direct measurements from indirect calorimetry.
Estimated Lower-Limb Muscle Activation Derived From Joint-Space Musculoskeletal Modeling | through study completion, an average of 1 year
  Lower-limb muscle activation patterns will be estimated using joint-space musculoskeletal models based on motion capture and ground reaction force data collected during treadmill walking. Estimated muscle activation values will be computed on a stride-by-stride basis to characterize neuromuscular engagement during exoskeleton-assisted gait.
Lower-Limb Muscle Activation Measured by Surface Electromyography During Walking | through study completion, an average of 1 year
  Muscle activation of lower-limb muscles (e.g., tibialis anterior, gastrocnemius medialis, gastrocnemius lateralis, soleus) will be measured during treadmill walking using surface electromyography (Delsys). EMG signals will be collected continuously and processed to quantify muscle activation patterns during exoskeleton-assisted gait.
During treadmill walking trials conducted at a single study visit | through study completion, an average of 1 year
  Controller parameter convergence will be assessed during human-in-the-loop optimization trials by evaluating changes in controller gain and timing parameters across successive walking bouts. Convergence is defined as stabilization of controller parameters within a predefined range during the optimization process.

CONTACTS AND LOCATIONS:
Overall Officials: Farah Fallahtafti, PhD, Principal Investigator — Department of Biomechanics, University of Nebraska at Omaha
Locations (1):
- Biomechanics Research Building, University of Nebraska at Omaha, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because direct measurements are only taken for baseline measurements that the modeling software will be using. The scripts and code used will be shared through opensource, but that does not include subject data.